CLINICAL TRIAL: NCT04869358
Title: Tracking the Immune Response to SARS-CoV-2 modRNA Vaccines in an Open-label Multicenter Study in Participants With Relapsing Multiple Sclerosis Treated With Ofatumumab s.c. (KYRIOS)
Brief Title: Exploring the Immune Response to SARS-CoV-2 COVID-19 Vaccines in Patients With Relapsing Multiple Sclerosis (RMS) Treated With Ofatumumab
Acronym: KYRIOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GDE01
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: COVID-19; SARS-CoV-2 mRNA vaccine; immune response; Ofatumumab; Relapsing Multiple Sclerosis; RMS; adult; MS
MeSH Terms: conditions — COVID-19 | interventions — ofatumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1a (Experimental): Patients received first SARS-CoV-2 vaccination within the study prior to starting ofatumumab treatment.
  Interventions: Drug: Ofatumumab
- Cohort 1b (Experimental): Patients had already completed initial vaccination cycle and received a booster vaccine within the study prior to starting ofatumumab treatment.
  Interventions: Drug: Ofatumumab
- Cohort 2a (Experimental): Patients who received their first SARS-CoV-2 vaccination within the study while already stable on ofatumumab treatment for at least 4 weeks (since the first dose).
  Interventions: Drug: Ofatumumab
- Cohort 2b (Experimental): Patients who had already completed their initial vaccination cycle and received a booster vaccine within the study while already stable on ofatumumab treatment for at least 4 weeks (since the first dose).
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab 20 mg s.c. on days 1, 7, 14, week 4 and every 4 weeks thereafter
  Other Names: OMB157

SUMMARY:
This study aimed to understand whether patients with relapsing multiple sclerosis (RMS) can mount an immune response to SARS-CoV-2 mRNA vaccines (initial vaccinations or booster vaccines) when vaccinated either before initiation of ofatumumab treatment or at least 4 weeks after commencing ofatumumab treatment.

DETAILED DESCRIPTION:
This was a four cohort, multicenter, open-label, prospective study of 34 (optionally up to 60) patients who had relapsing multiple sclerosis (RMS) planning to undergo a SARS-CoV-2 mRNA vaccination (initial vaccinations or booster vaccines) as part of clinical routine. The maximal duration of the study for an individual patient was 22 months.

* The first cohort was RMS patients receiving SARS-CoV-2 mRNA vaccine (initial vaccinations or booster vaccines) as part of clinical routine prior to starting ofatumumab treatment.
* The second cohort was participants receiving SARS-CoV-2 mRNA vaccine (initial vaccinations or booster vaccines) as part of clinical routine while already stable on ofatumumab treatment for at least 4 weeks (since first dose).

Cohort 1a - Patients received first SARS-CoV-2 vaccination within the study prior to starting ofatumumab treatment.

Cohort 1b - Patients had already completed initial vaccination cycle and received a booster vaccine within the study prior to starting ofatumumab treatment.

Cohort 2a - Patients who received their first SARS-CoV-2 vaccination within the study while already stable on ofatumumab treatment for at least 4 weeks (since the first dose).

Cohort 2b - Patients who had already completed their initial vaccination cycle and received a booster vaccine within the study while already stable on ofatumumab treatment for at least 4 weeks (since the first dose).

Development of SARS-CoV-2 specific T-cells and functional anti-SARS-CoV-2 antibodies were investigated for up to 18 months after the participants' vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Multiple Sclerosis (RMS) diagnosis
* eligible for ofatumumab treatment
* willing and eligible to receive SARS-CoV-2 mRNA vaccine

Exclusion Criteria:

* known prior or current COVID-19 infection
* previous treatment with BTK inhibitor or anti-CD20 therapy other than ofatumumab
* no previous vaccination with a non-modRNA SARS-CoV-2 vaccine.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Unterhaching

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2143

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-seven participants were screened and 34 participants met the criteria for entry into the trial.
Period: Overall Study
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b
Started | 6 | 8 | 5 | 15
Completed | 5 | 8 | 5 | 15
Not Completed | 1 | 0 | 0 | 0
Not completed — Wish to have children. | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Total
Number analyzed (Participants) | 6 | 8 | 5 | 15 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.1) | 47.1 (14.1) | 32.4 (7.7) | 45.5 (12.4) | 41.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 9 | 23
  Male | 1 | 3 | 1 | 6 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 6 | 8 | 5 | 13 | 32
  Missing | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Having Established SARS-CoV-2-specific T Cells After Receiving a modRNA Vaccine
Description: Participants who established SARS-CoV-2-specific T cells as defined by detection of SARS-CoV-2 reactive T-cells, measured by e.g. ELIspot assay from T-cells that were stimulated with SARS-CoV-2 peptide mix, either 1 month after second dose of vaccine or 1 month after booster vaccine in participants who received the respective vaccine before or after starting ofatumumab treatment.
Time Frame: 1 month after second dose of vaccine or booster vaccine
Population: Efficacy and safety analysis sets
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: All cohorts
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Total
Number analyzed (Participants) | 5 | 8 | 4 | 15 | 32
percentage of participants | 80.0 [28.4 to 99.5] | 87.5 [47.3 to 99.7] | 100.0 [39.8 to 100.0] | 46.7 [21.3 to 73.4] | 68.8 [50 to 83.9]

2. Secondary Outcome: Percentage of Participants Who Maintained T-cell Response After Receiving a modRNA Vaccine
Description: Participants who maintained detectable SARS-CoV-2 reactive T-cells (measured by e.g. ELIspot assay from T-cells that were stimulated with SARS-CoV-2 peptide mix) after second dose of vaccine or 6 and 12 months after booster vaccine in participants who received the vaccine before or after starting ofatumumab treatment. First booster vaccination was optional for cohorts 1a and 2a. In cohorts 1b and 2b the time points "Month 1 after Vacc" and "1 Month after booster" are identical.
Time Frame: At Week 1, Months 6, 12 and 18 after second dose of vaccine or 1 Month after 1st booster, 1 Month after 2nd booster
Population: Efficacy and safety analysis sets
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Total
Number analyzed (Participants) | 6 | 8 | 5 | 15 | 34
percentage of participants
  Week 1 after vacc n=4,0,5,0,9: number analyzed (Participants) | 4 | 0 | 5 | 0 | 9
  Week 1 after vacc n=4,0,5,0,9 | 100.0 [39.8 to 100.0] |  | 100.0 [47.8 to 100.0] |  | 100.0 [66.4 to 100.0]
  Month 6 after vacc n=4,8,5,14,31: number analyzed (Participants) | 4 | 8 | 5 | 14 | 31
  Month 6 after vacc n=4,8,5,14,31 | 100 [39.8 to 100.0] | 62.5 [24.5 to 91.5] | 60.0 [14.7 to 94.7] | 57.1 [28.9 to 82.3] | 64.5 [45.4 to 80.8]
  Month 12 after vacc n=5,5,5,15,30: number analyzed (Participants) | 5 | 5 | 5 | 15 | 30
  Month 12 after vacc n=5,5,5,15,30 | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 80.0 [28.4 to 99.5] | 93.3 [68.1 to 99.8] | 93.3 [77.9 to 99.2]
  Month 18 after vacc n=4,0,4,0,8: number analyzed (Participants) | 4 | 0 | 4 | 0 | 8
  Month 18 after vacc n=4,0,4,0,8 | 50.0 [6.76 to 93.2] |  | 100.0 [39.8 to 100.0] |  | 93.3 [77.9 to 99.2]
  Month 1 after 1st booster n=4,8,3,15,30: number analyzed (Participants) | 4 | 8 | 3 | 15 | 30
  Month 1 after 1st booster n=4,8,3,15,30 | 75.0 [19.4 to 99.4] | 87.5 [47.3 to 99.7] | 66.7 [9.43 to 99.2] | 46.7 [21.3 to 73.4] | 63.3 [43.9 to 80.1]
  Month 1 after 2nd booster n=2,4,0,10,16: number analyzed (Participants) | 2 | 4 | 0 | 10 | 16
  Month 1 after 2nd booster n=2,4,0,10,16 | 100.0 [15.8 to 100.0] | 75.0 [19.4 to 99.4] |  | 80.0 [44.4 to 97.5] | 81.3 [54.4 to 96.0]

3. Secondary Outcome: Increase in Specific T-cells After Receiving an modRNA Booster Vaccine
Description: Patients having established SARS-CoV-2-specific T cells as defined by detection of SARS-CoV-2 reactive T-cells, measured by e.g. ELIspot assay from T-cells that were stimulated with SARS-CoV-2 peptide mix 1 month after booster vaccine in participants who received the respective vaccine before or after starting ofatumumab treatment. The fold change of SI from last value before booster to Month 1 is the ratio of SI at Month 1 divided by SI at last value before booster.
Time Frame: Last value before booster to 1 month after booster
Population: All patients in the efficacy analysis set, for whom ELISpot data for the time points "last visit before booster" and "month 1 after booster" were available, were included in the analysis.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Total
Number analyzed (Participants) | 4 | 7 | 3 | 14 | 28
fold change | 0.8 (0.9) | 12.6 (25.5) | 2.0 (2.1) | 3.6 (4.4) | 5.3 (13.2)

4. Secondary Outcome: Percentage of RMS Participants With Quantifiable Levels of SARS-CoV-2 Serum Functional Antibodies by Visits and Subcohorts (EAS)
Description: Level of SARS-CoV-2 serum functional antibodies were measured by a central laboratory using a neutralizing antibody detection kit.
Time Frame: Baseline, Week 1 after Vacc, Month 1, 6, 12 after Vacc, 1 month after 1st booster, 1 month after 2nd booster
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b
Number analyzed (Participants) | 6 | 8 | 5 | 15
percentage of participants
  Baseline0 positive n=6,8, 5,14: number analyzed (Participants) | 6 | 8 | 5 | 14
  Baseline0 positive n=6,8, 5,14 | 0 [0 to 45.9] | 100.0 [63.1 to 100.0] | 0 [0 to 52.2] | 71.4 [41.9 to 91.6]
  Week 1 after Vacc positive n=5,0,5,0: number analyzed (Participants) | 5 | 0 | 5 | 0
  Week 1 after Vacc positive n=5,0,5,0 | 100.0 [47.8 to 100.0] |  | 40.0 [5.27 to 85.3] |
  Month 1 after Vacc positive n=5,8,4,15: number analyzed (Participants) | 5 | 8 | 4 | 15
  Month 1 after Vacc positive n=5,8,4,15 | 100.0 [47.8 to 100.0] | 100.0 [63.1 to 100.0] | 25.0 [0.63 to 80.6] | 93.3 [68.1 to 99.8]
  Month 6 after Vacc positive n=5,8,5,15: number analyzed (Participants) | 5 | 8 | 5 | 15
  Month 6 after Vacc positive n=5,8,5,15 | 100.0 [47.8 to 100.0] | 100.0 [63.1 to 100.0] | 40.0 [5.3 to 85.3] | 73.3 [44.9 to 92.2]
  Month 12 after Vacc positive n=5,7,5,14: number analyzed (Participants) | 5 | 7 | 5 | 14
  Month 12 after Vacc positive n=5,7,5,14 | 100.0 [47.8 to 100.0] | 100.0 [59.0 to 100.0] | 40.0 [5.3 to 85.3] | 92.9 [66.1 to 99.8]
  Month 1 after 1st booster postive n=5,8,5,15: number analyzed (Participants) | 5 | 8 | 5 | 15
  Month 1 after 1st booster postive n=5,8,5,15 | 100.0 [47.8 to 100.0] | 100.0 [63.1 to 100.0] | 66.7 [9.4 to 99.2] | 93.3 [68.1 to 99.8]
  Month 1 after 2nd booster positive n=2,4,0,10: number analyzed (Participants) | 2 | 4 | 0 | 10
  Month 1 after 2nd booster positive n=2,4,0,10 | 100.0 [15.8 to 100.0] | 100.0 [39.8 to 100.0] |  | 90.0 [55.5 to 99.7]

5. Secondary Outcome: SARS-CoV-2 Specific CD4+ Effector Memory T-cells
Description: Phenotypic description of the cellular immune response was performed at the central laboratory. T-cells were stimulated with SARS-CoV-2 peptide mix and analyzed for IFNg- and IL4 secretion using FACS analysis.
Time Frame: Baseline, Months 1 ,6, 12 and 18 after vaccinationse of vaccine or 1,6 and 12 months after booster vaccine
Population: Full analysis set -available participant data varied across time points. In alignment with the secondary study objectives of the protocol and the corresponding statistical analysis plan, the phenotypical parameters were assessed by cohort. Therefore, participants in the subcohorts 1a/1b and 2a/2b were combined.
Measure: Mean (Standard Deviation); unit: % of CD4+/CD8+ cells
Groups:
- Cohort 1: Patients received SARS-CoV-2 vaccination (initial or booster) within the study prior to starting ofatumumab treatment.
- Cohort 2: Patients received SARS-CoV-2 vaccination (initial or booster) within the study while already stable on ofatumumab treatment for at least 4 weeks (since the first dose).
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 14 | 20
% of CD4+/CD8+ cells
  BL before initial Vacc IL4 basal n=4,5: number analyzed (Participants) | 4 | 5
  BL before initial Vacc IL4 basal n=4,5 | 2.458 (4.915) | 0.262 (05.86)
  BL before initial Vacc IL4 stim.n=4,5: number analyzed (Participants) | 4 | 5
  BL before initial Vacc IL4 stim.n=4,5 | 2.583 (5.165) | 0.264 (0.59)
  BL before initial Vacc INFg basal n=4,5: number analyzed (Participants) | 4 | 5
  BL before initial Vacc INFg basal n=4,5 | 0.555 (0.549) | 0.03 (0.067)
  BL before initial Vacc INGg stim n=4,5: number analyzed (Participants) | 4 | 5
  BL before initial Vacc INGg stim n=4,5 | 0.235 (0.191) | 0.146 (0.326)
  Month 1 after Vacc Il4 basal n=12,19: number analyzed (Participants) | 12 | 19
  Month 1 after Vacc Il4 basal n=12,19 | 0.396 (2.318) | 1.209 (6.919)
  Month 1 after Vacc IL4 stim. n=12,19: number analyzed (Participants) | 12 | 19
  Month 1 after Vacc IL4 stim. n=12,19 | 0.719 (0.62) | 2.449 (0.283)
  Month 1 after Vacc INFg basal n=12,19: number analyzed (Participants) | 12 | 19
  Month 1 after Vacc INFg basal n=12,19 | 0.258 (2.165) | 0.171 (0.917)
  Month 1 after Vacc INFg stim. n=12,19: number analyzed (Participants) | 12 | 19
  Month 1 after Vacc INFg stim. n=12,19 | 0.947 (2.165) | 0.381 (0.917)
  Month 6 after Vacc Il4 basal n=12,20: number analyzed (Participants) | 12 | 20
  Month 6 after Vacc Il4 basal n=12,20 | 0.662 (1.44) | 0.061 (0.273)
  0Month 6 after Vacc IL4 stim.n=12,20: number analyzed (Participants) | 12 | 20
  0Month 6 after Vacc IL4 stim.n=12,20 | 0.93 (2.043) | 0.44 (0.197)
  Month 6 after Vacc INFg basal n=12,20: number analyzed (Participants) | 12 | 20
  Month 6 after Vacc INFg basal n=12,20 | 0.236 (0.344) | 0.123 (0.205)
  Month 6 after Vacc INFg stim.n=12,20: number analyzed (Participants) | 12 | 20
  Month 6 after Vacc INFg stim.n=12,20 | 0.305 (0.352) | 0.342 (0.644)
  Month 12 after Vacc Il4 basal n=10,17: number analyzed (Participants) | 10 | 17
  Month 12 after Vacc Il4 basal n=10,17 | 0.361 (1.142) | 1.078 (2.468)
  Month 12 after Vacc IL4 stim.n=10,17: number analyzed (Participants) | 10 | 17
  Month 12 after Vacc IL4 stim.n=10,17 | 0.174 (0.55) | 1.031 (2.491)
  Month 12 after Vacc INFg basal n=10,17: number analyzed (Participants) | 10 | 17
  Month 12 after Vacc INFg basal n=10,17 | 0.132 (0.192) | 0.226 (0.478)
  Month12 after Vacc INFg stim. n=10,17: number analyzed (Participants) | 10 | 17
  Month12 after Vacc INFg stim. n=10,17 | 0.122 (0.26) | 0.757 (2.332)
  Month 18 after Vacc IL4 basal n=4,5: number analyzed (Participants) | 4 | 5
  Month 18 after Vacc IL4 basal n=4,5 | 2.368 (4.735) | 0.118 (0.264)
  Month 18 after Vacc IL4 stim.l n=4,5: number analyzed (Participants) | 4 | 5
  Month 18 after Vacc IL4 stim.l n=4,5 | 1.833 (3.665) | 0.176 (0.394)
  Month 18 after Vacc INFg basal l n=4,5: number analyzed (Participants) | 4 | 5
  Month 18 after Vacc INFg basal l n=4,5 | 0.148 (0.295) | 0.11 (0.246)
  Month 18 after Vacc INFg stim.l n=4,5: number analyzed (Participants) | 4 | 5
  Month 18 after Vacc INFg stim.l n=4,5 | 0.138 (0.159) | 0.12 (0.268)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until the end of the treatment period plus an additional 30 day safety follow up period for a maximum time of 22 months.
Groups:
- Cohort 1b: Patients had already completed initial vaccination cycle and received a booster vaccine within the study prior to starting ofatumumab treatmen
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 1/5 | 1/15
Other Adverse Events (participants affected / at risk) | 6/6 | 6/8 | 5/5 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=6) | Cohort 1b (N=8) | Cohort 2a (N=5) | Cohort 2b (N=15)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=6) | Cohort 1b (N=8) | Cohort 2a (N=5) | Cohort 2b (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 3 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 0
Immune-mediated adverse reaction (Immune system disorders) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 2 | 5 | 9
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 3
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 4 | 3
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 1 | 1 | 0
Peripheral nerve lesion (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Immunophenotyping (outcome measure 5) was inconclusive due to low participant numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04869358/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT04869358/SAP_001.pdf